CLINICAL TRIAL: NCT01185223
Title: Multicenter, Randomized Study Comparing Oral Valganciclovir Versus Intravenous Ganciclovir in Patients Following Allogeneic Stem Cell Transplantation
Brief Title: Study Comparing Valganciclovir Versus Ganciclovir in Patients Following Allogeneic Stem Cell Transplantation
Acronym: CONVINCE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pierrel Research Europe GmbH (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Pierrel Research Europe GmbH, Pierrel Research Europe GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ML 22371
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Allogeneic Stem Cell Transplantation
Keywords: Valganciclovir; Ganciclovir; Antiviral Drug; CMV disease
MeSH Terms: conditions — Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Valganciclovir; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valganciclovir (Other)
  Interventions: Drug: Valganciclovir
- Ganciclovir (Active Comparator)
  Interventions: Drug: Ganciclovir

INTERVENTIONS:
Drug: Valganciclovir — Valganciclovir 450mg tablet or Valganciclovir powder for oral solution 50mg/mL
  Other Names: Ro 107-9070; Valcyte
  Arms: Valganciclovir
Drug: Ganciclovir — 2x5mg/kg/d intravenous ganciclovir
  Other Names: Cymeven
  Arms: Ganciclovir

SUMMARY:
The objective of this study is to assess the efficacy and safety of oral valganciclovir versus intravenous ganciclovir in patients following allogenic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient following allogeneic SCT
* Patient with a first episode of positive CMV-PCR (DNAemia) or pp65 antigenemia assay (antigenemia) up to 100 days after SCT
* Absolute neutrophil count (ANC) ≥1000 cells/µL on 2 consecutive follow-ups within 10 days before randomization
* Patient has a creatinine clearance of ≥25 mL/min (calculated by the Cockcroft-Gault formula, see Part I Section 6.1.2) with evidence of improving renal function,
* None or gastrointestinal graft-versus-host disease (GVHD) up to grade 2

Exclusion Criteria:

* Patient has a suspected or diagnosed CMV disease
* Patient has received syngeneic SCT
* Patient who received an investigational medicinal product (IMP) within the last 30 days prior to screening or who is simultaneously participating in another clinical study with an IMP
* Patient with a body weight <50 kg or >95 kg,
* Patient has received anti-CMV therapy within the past 30 days prior to screening (the use of acyclovir, valacyclovir, or famciclovir is permitted)
* Patient who has participated in this study before,
* Patient who shows a neutropenia, thrombocytopenia, or anemia within 10 days before or at the time point of randomization as following:

  * The ANC is <1000 cells/μL on 2 consecutive follow-ups, or
  * A platelet count of ≥25000/μL can not be achieved/maintained with platelet transfusions
  * A hemoglobin level of ≥8g/dL can not be achieved/maintained by red blood cell transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy and Safety of oral valganciclovir versus intravenous ganciclovir | max. 2 years (recruitement time)
  Main variable for efficacy in the primary endpoint will be evaluated by assessment of the event-free survival within 180 days after stem cell transplantation.
  Main variable for safety in the primary endpoint will be evaluated by the porpotion of patients with severe neutropenia until 7 days after discontinuation of antiviral therapy with the study drug.

SECONDARY OUTCOMES:
Combined secondary endpoint of efficacy and safety | max. 2 years (recruitement time)
  The secondary variables of efficacy will be:
  The proportion of patients with persistently positive blood specimens for CMV after completion of antiviral therapy with the Study Drug,
  * The proportion of patients who require retreatment after discontinuation of antiviral therapy with the Study Drug until day 180,
  * The proportion of patients with CMV disease within 180 days after SCT,
  * The number of days patients were alive and not hospitalized between randomization and day 180 post SCT,
  * The proportion of patients who died from any cause within 180 days after SCT.

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Einsele, Prof. Dr., Principal Investigator — Hospital
Locations (17):
- Pierrel Site 50, Vienna, Austria
- Germany (10):
  - Pierrel Site 12, Berlin
  - Pierrel Site 13, Berlin
  - Pierrel Site 9, Bremen
  - Pierrel Site 3, Essen
  - Pierrel Site 7, Kiel
  - Pierrel Site 5, Leipzig
  - Pierrel Site 4, Münster
  - Pierrel Site 8, Oldenburg
  - Pierrel Site 10, Rostock
  - Pierrel Site 1, Würzburg
- Spain (6):
  - Pierrel Site 32, Barcelona
  - Pierrel Site33, Barcelona
  - Pierrel Site 30, Madrid
  - Pierrel Site 34, Madrid
  - Pierrel Site 31, Salamanca
  - Pierrel Site 35, Valencia